CLINICAL TRIAL: NCT04489654
Title: Evaluation of Immediate Implant Placement With a Modified Socket Shield Technique Using Xenogenic Bone Graft. (a Randomized Controlled Clinical Trial) CLINICAL TRIAL)
Brief Title: Immediate Implant Using Socket Shield Technique With Xenogenic Bone Graft
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: interventional
Record Dates: First submitted 2020-07-19; First posted 2020-07-28 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2019-07

CONDITIONS: Immediate Implant

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study (Active Comparator): Test group will receive immediate implant with modified socket shield and deproteinized bovine bone mineral (DBBM) OneXeno Graft. ( OneGraft, Germany) put in the buccal gap
  Interventions: Biological: deproteinized bovine bone mineral (DBBM) by OneXeno Graft. ( OneGraft, Germany)
- control (No Intervention): Control group will receive an immediate implant with modified socket shield technique but without deproteinized bovine bone mineral (DBBM) OneXeno Graft. ( OneGraft, Germany) in the buccal gap

INTERVENTIONS:
Biological: deproteinized bovine bone mineral (DBBM) by OneXeno Graft. ( OneGraft, Germany) — deproteinized bovine bone mineral (DBBM) put in the gap between implant and labial shield
  Arms: study

SUMMARY:
Adequate bone volume and a proper aesthetic outcome have become the main focus of interest in implant dentistry. Alveolar bone resorption is a natural course occurring after tooth removal. Partial extraction therapy through root preservation has been reported to help in bone maintenance at the extraction site. In 2010, Hurzeler et al. evaluated a new approach, at that time, called socket shield technique. Han et al. in 2018 reported the modification of this technique and leaving the jump gap between the shield and the implant non-grafted. The importance of bone grafting of the gap between the implant and the labial shield in improving quality of regenerating bone and prevention of the soft tissue ingrowth has been described. Thus the hypothesis, of improving the modified socket shield technique by bone grafting could be tested.

Aim of this study is to evaluate the clinical and radiographic outcomes of using xenogenic bone graft on outcome of immediate dental implant placement using the modified socket shield technique.

DETAILED DESCRIPTION:
16 patients who are admitted to the outpatient clinic of Oral and Maxillofacial Surgery Department, are divided into two study groups. Control group will receive an immediate implant with modified socket shield technique. Test group will receive immediate implant with modified socket shield and deproteinized bovine bone mineral (DBBM) put in the buccal gap. Outcome measurement is primary and secondary implant stability measurement and CBCT evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Age more than 18 years old irrespective of the gender
* One or more of non-restorable (fractured or decayed) tooth/teeth in the upper aesthetic regions (incisors, premolars).
* Free from periodontal diseases.
* Sufficient bone volume to allow placement of an implant.
* Ability to read and sign an informed consent form
* Adequate buccolingual width to allow for a buccal gap presence.

Exclusion Criteria:

* A medical history that contraindicates oral surgical treatment (uncontrolled/untreated diabetes mellitus, immuno-compromised status, radio/chemotherapy of the oral and maxillofacial region, treatment with oral and/or intravenous amino-bisphosphonates).
* Untreated periodontal disease.
* Vertical root fractures on the buccal aspect.
* Tooth /teeth with horizontal fractures below bone level.
* Tooth /teeth with external or internal resorptions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2019-07-20 (Actual); Primary Completion 2020-08-14 (Estimated); Study Completion 2020-10-01 (Estimated)

PRIMARY OUTCOMES:
primary and secondary implant stability measurement | 4 months
  Implant stability measured in units ISQ is concluded through a clinical evaluation using ostell

SECONDARY OUTCOMES:
Bone mineral density | 6 months
  Bone mineral density is calculated through radiographic evaluation by means of cone beam CT

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandra university, Alexandria, Egypt